CLINICAL TRIAL: NCT03895684
Title: Phase 1 Trial of the LSD1 Inhibitor SP-2577 (Seclidemstat) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Salarius Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SALA-003-AC19
Record Dates: First submitted 2019-02-14; First posted 2019-03-29 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: This single arm study will utilize an accelerated dose escalation, followed by a conventional 3+3 dose escalation phase to achieve maximum tolerated dose (MTD).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sp-2577 (Experimental): Twice-daily administration of oral SP-2577
  Interventions: Drug: SP-2577 Seclidemstat

INTERVENTIONS:
Drug: SP-2577 Seclidemstat — Dose escalation and dose expansion of SP-2577.
  Other Names: LSD1 Inhibitor

SUMMARY:
Phase 1, open-label, non-randomized dose finding study of SP-2577 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Phase 1, open-label, non-randomized dose finding study of SP-2577 given as oral tablets in patients with advanced solid tumors in 28-day cycles. The study design is based on a Simon's 4B design without intrapatient dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years and weight ≥ 40 kg.
* Diagnosis of advanced or recurrent, histologically or cytologically confirmed, solid malignancy that is either metastatic or unresectable. At time of enrollment, subjects must have progressed on, be intolerant of, refuse, or ineligible for, all available standard of care therapies.
* Subjects must demonstrate measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, with the exception of castration-resistant prostate cancer (CRPC) who should have progression based on the PCWG 3.0 criteria
* Karnofsky ≥70% for over ≥16 years old and Lansky ≥70% for under 16 years old, equivalent to Eastern Cooperative Oncology Group (ECOG) performance status grade 0 or 1
* Willingness to provide tumor biopsies of assessible lesions on and off treatment (Dose expansion cohort only). Optional for patients <18 years of age.
* Able to swallow and retain orally administered medication.
* Patients must have normal organ and marrow function
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects with Ewing Sarcoma. See NCT03600649, Protocol Number: SALA-002-EW16.
* Subjects with primary central nervous system tumors
* Patients who have not recovered to grade 1 or baseline from adverse events related to prior therapy excluding lymphopenia, alopecia, peripheral neuropathy and ototoxicity, which are excluded if ≥ CTCAE grade 3 (Version 5.0).
* Patients who are receiving any other investigational agents.
* Prior therapy with LSD1 targeted agents including monoamine oxidases for cancer therapy.
* Prior systemic anti-cancer treatment (chemotherapy, biologic therapy [ie. small molecular inhibitors, monoclonal antibodies]) within 21 days prior to Cycle 1 Day 1.
* Prior therapy with immunotherapy such as a checkpoint inhibitor, cellular therapy or vaccine therapy within 28 days prior to Cycle 1 Day 1. Patients must have recovered from any immune-related adverse events to grade 1 or baseline and require ≤ 10 mg of prednisone equivalents daily. Patients with immune-related hypothyroidism and/or hypoadrenalism may enroll while on thyroid or hydrocortisone replacement therapy, respectively.
* Prior small port palliative radiotherapy within 14 days or 42 days from definitive local control radiation (any dose greater than 50Gy).
* Anti-androgen therapies for prostate cancer, such as bicalutamide, within 4 weeks prior to enrollment. Second-line hormone therapies such as enzalutamide, abiraterone, or orteronel within 2 weeks prior to enrolment. Subjects with prostate cancer should remain on luteinizing hormone releasing hormone (LHRH) agonists or antagonists. Subjects with prostate cancer may also remain on low-dose prednisone or prednisolone up to 10 mg/day
* Prior therapy with long acting myeloid growth factor within 14 days or 7 days from a short acting myeloid growth factor.
* Participation in a prior investigational study within 30 days prior to Cycle 1 Day 1.
* Patients with progressive or symptomatic brain metastases. Patients with brain metastases may be included in this trial as long as the brain metastases have received definitive treatment and are stable (i.e., no evidence of progression). The brain metastases must be stable for a minimum of 6 weeks.
* Patients must have discontinued anti-seizure medications and steroids, except for physiologic steroid dosing (≤10 mg/day of prednisone equivalents).
* Patients currently receiving any of the following substances and cannot be discontinued 14 days prior to Cycle 1 Day 1: Moderate or strong inhibitors or inducers of major CYP isoenzymes, including grapefruit, grapefruit hybrids, pomelos, star-fruit, and Seville oranges; Moderate or strong inhibitors or inducers of major drug transporters; Substrates of CYP3A4/5 with a narrow therapeutic index
* Uncontrolled concurrent illness including, but not limited to: ongoing or active infection; transfusion dependent thrombocytopenia or anemia; psychiatric illness/social situations that would limit compliance with study requirements
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following: symptomatic congestive heart failure; Left Ventricular Ejection Fraction (LVEF) ≤ 50%; unstable angina pectoris or cardiac arrhythmia; baseline QTcF (Fridericia) ≥ 450 milliseconds; Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome
* Any major surgery within 21 days prior to Cycle 1 Day 1.
* Pregnant and breastfeeding women
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with SP-2577. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SP-2577 | From screening through at least 30 days after end of treatment, up to approximately 24 months
  Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0

SECONDARY OUTCOMES:
Determine the maximum tolerated dose of SP-2577 | DLTs within the first cycle of therapy (up to 28 days)
  Defined as the dose level immediately below the dose level at which ≥ 2 patients from a cohort of 3 to 6 patients experience a dose-limiting toxicity (DLT).
Characterization of pharmacokinetics of SP-2577 (area under the concentration time profile) | At protocol defined time points on cycle 1 (each cycle is 28 days), day 1 and 2 and cycle 2, day 1 and 2.
  SP-2577 under fasted and fed conditions
Characterization of pharmacokinetics of SP-2577 (time to maximum plasma concentration) | At protocol defined time points on cycle 1 (each cycle is 28 days), day 1 and 2 and cycle 2, day 1 and 2.
  SP-2577 under fasted and fed conditions
Characterization of pharmacokinetics of SP-2577 (maximum plasma concentration) | At protocol defined time points on cycle 1 (each cycle is 28 days), day 1 and 2 and cycle 2, day 1 and 2.
  SP-2577 under fasted and fed conditions
Characterization of pharmacokinetics of SP-2577 (half-life) | At protocol defined time points on cycle 1 (each cycle is 28 days), day 1 and 2 and cycle 2, day 1 and 2.
  SP-2577 under fasted and fed conditions
Characterization of pharmacokinetics of SP-2577 (clearance rate) | At protocol defined time points on cycle 1 (each cycle is 28 days), day 1 and 2 and cycle 2, day 1 and 2.
  SP-2577 under fasted and fed conditions
Characterization of pharmacokinetics of SP-2577 (volume of distribution) | At protocol defined time points on cycle 1 (each cycle is 28 days), day 1 and 2 and cycle 2, day 1 and 2.
  SP-2577 under fasted and fed conditions
Efficacy parameter: overall response rate of SP-2577 | From start of treatment through at least 30 days after end of treatment, up to approximately 24 months
  Assessed by radiographic imaging with response and progression evaluated by RECIST 1.1 guidelines
Efficacy parameter: duration of response of SP-2577 | From start of treatment through at least 30 days after end of treatment, up to approximately 24 months
  Assessed by radiographic imaging with response and progression evaluated by RECIST 1.1 guidelines
Efficacy parameter: progression-free survival of SP-2577 | From start of treatment through at least 30 days after end of treatment, up to approximately 24 months
  Assessed by radiographic imaging with response and progression evaluated by RECIST 1.1 guidelines
Changes in serum hemoglobin F concentrations | At protocol defined time points from start of treatment through end of treatment, up to approximately 24 months
  Determine changes serum hemoglobin F concentrations correlated with SP-2577 treatment and clinical and radiographic markers of disease burden (either response or resistance/progression).
Changes in the molecular signatures of the tumor | At protocol defined time points from start of treatment through end of treatment, up to approximately 24 months
  Assessed in dose expansion only by RNA-seq testing of tumor biopsy samples to determine changes in gene expression patterns by SP-2577 treatment to elucidate biological changes induced in the tumor by LSD1 inhibition.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - HonorHealth, Scottsdale, Arizona
  - Sarcoma Oncology Research Center, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No